CLINICAL TRIAL: NCT06437977
Title: Neoadjuvant Therapy of SBRT Sequencial with Toripalimab and Chemotherapy in Resectable Stage II-III NSCLC Patients: a Multicenter, Openlabel, Randomized, Phase III Trial
Brief Title: Neoadjuvant Therapy of SBRT Sequencial with Toripalimab and Chemotherapy in Resectable Stage II-III NSCLC Patients(neoR-TORCH)
Acronym: neoR-TORCH
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Xuwei Cai, Director, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IS24056
Record Dates: First submitted 2024-05-26; First posted 2024-05-31 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Stage II-III Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — toripalimab

STUDY DESIGN:
Intervention Model Description: Parallel
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): Participants receive SBRT for primary lung tumor, sequential receive totally 4 cycles of Toripalimab combined with platinum doublet chemotherapy during perioperative period ; participants receive consolidation therapy of Toripalimab Intervention: SBRT: 24Gy/3fractions; Drug: 4cycles(Toripalimab IV 240mg + platinum-based doublet chemotherapy)+13 cycles(Toripalimab IV 240mg); Biological: Toripalimab
  Interventions: Radiation: SBRT; Drug: Toripalimab
- Active Comparator (Active Comparator): Participantsreceive totally 4 cycles of Toripalimab combined with platinum doublet chemotherapy during perioperative period ; participants receive consolidation therapy of Toripalimab Intervention: Drug: 4cycles(Toripalimab IV 240mg + platinum-based doublet chemotherapy)+13 cycles(Toripalimab IV 240mg); Biological: Toripalimab
  Interventions: Drug: Toripalimab

INTERVENTIONS:
Radiation: SBRT — SBRT. 24Gy/3fractions Toripalimab 240 mg by IV infusion every 3 weeks (Q3W), given on cycle day 1;Drug: Cisplatin 75 mg/m^2 by IV infusion Q3W, given on cycle day 1;Drug: Corboplatin AUC 5 by IV infusion Q3W, given on cycle day 1;Drug: Pemetrexed 500 mg/m^2 by IV infusion Q3W, given on cycle day 1. Given only to participants with nonsquamous NSCLC.Drug:Paclitaxel 175 mg/m^2 by IV infusion Q3W;Drug:Docetaxel 60-75 mg/m^2 by IV infusion Q3W
  Arms: Experimental
Drug: Toripalimab — Toripalimab 240 mg by IV infusion every 3 weeks (Q3W), given on cycle day 1;Drug: Cisplatin 75 mg/m^2 by IV infusion Q3W, given on cycle day 1;Drug: Corboplatin AUC 5 by IV infusion Q3W, given on cycle day 1;Drug: Pemetrexed 500 mg/m^2 by IV infusion Q3W, given on cycle day 1. Given only to participants with nonsquamous NSCLC.Drug:Paclitaxel 175 mg/m^2 by IV infusion Q3W;Drug:Docetaxel 60-75 mg/m^2 by IV infusion Q3W
  Other Names: Toripalimab IV 240mg + platinum-based doublet chemotherapy

SUMMARY:
This is a randomized, controlled, multi-center, phase III clinical study to evaluate the efficacy and safety of SBRT sequencial with Toripalimab and chemotherapy versus Toripalimab and chemotherapy for subjects with resectable, stage II-III NSCLC.

DETAILED DESCRIPTION:
Subjects who meet all the inclusion criteria but do not meet any exclusion criteria are randomized into two groups at a ratio of 1:1: according to the stratification factors as below:

* Disease stage: II vs IIIA vs IIIB
* PD-L1 status: PD-L1 expression ≥1% vs. PD-L1 <1% or not evaluable
* Pathological type: non-squamous cell carcinoma vs. squamous cell carcinoma Neoadjuvant therapy should be started within 1 week after randomization. Stereotactic body radiation therapy (SBRT) will be given for primary lung tumor, 24Gy/3fractions, sequential toripalimab IV 240 mg Q3W will be given combined with platinum-based doublet drug chemotherapy for three cycles in the preoperative neoadjuvant therapy period for trial group; the controlled group receive toripalimab IV 240 mg Q3W combined with platinum-based doublet drug chemotherapy for three cycles in the preoperative neoadjuvant therapy period. Every 3 weeks of treatment is regarded as one cycle, in which combined therapy is given in the first day of every cycle.

All the subjects will receive preoperative radiological and surgical evaluation 4-6 weeks after neoadjuvant therapy.

After 3 cycles of preoperative neoadjuvant therapy, all the subjects who still have surgical indications will receive radical excision based on the surgical operation criteria of the World Association for Lung Cancer Research within 4-6 weeks after 3 cycles of preoperative neoadjuvant therapy. The pTNM will be staged in accordance with AJCC Cancer Staging Manual (version 8). All the specimens taken during the operation will be evaluated by local pathologists for the surgical margin. The tumor tissue samples collected from subjects during the study will be submitted to the authorized central laboratory for blinded evaluation of pathological response and translational research.

All the subjects who have completed the radical operation will receive one cycle of postoperative adjuvant therapy, i.e., Toripalimab IV 240 mg/placebo + platinum-based doublet drug chemotherapy in 30 days after the operation. Then it will proceed to consolidation treatment period three weeks after adjuvant therapy; In the consolidation treatment period, Toripalimab IV 240 mg/placebo is given in each cycle of every 3 weeks for a total of 13 cycles . Adverse events (AEs) will be monitored throughout the study, and the severity will be graded to the guidelines listed in National Cancer Institute (NCI) common terminology criteria for adverse events (CTCAE) version 5.0 or above. The safety will be followed up in the subjects who have received study treatment and discontinued the drug prematurely. All the subjects will be followed up for overall survival, until death, withdrawal of informed consent or end of study

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 -75 years, regardless of gender；
2. ECOG score 0-1;
3. Treatment-naive, histologically confirmed resectable, stage II, IIIA, IIIB (N2) (AJCC staging system, version 8) NSCLC ;
4. Measurable lesions based on the response evaluation criteria in solid tumors version 1.1;
5. Tumor tissue specimens available for pathological diagnosis, detection of PD-L1 expression and biomarkers prior to randomization ;
6. According to the doctor's judgment, lung function can meet the requirements of pneumonectomy;
7. Confirming the absence of EGFR/ALK sensitive gene mutations through molecular pathological diagnosis of the organization;
8. Good organ function:

   Bone marrow function: absolute neutrophil count ≥ 1.5 × 109/L, platelet count ≥ 80 × 109/L, hemoglobin ≥9 g/dL; Liver function: total bilirubin ≤ 1.5 × ULN, ALT and AST ≤ 1.5 × ULN; Renal function: serum creatinine ≤ 1.5 × ULN or serum creatinine clearance rate ≥ 60 mL/min; blood urea nitrogen ≤ 200mg/L;
9. Having sufficient understanding of this study and being willing to sign the informed consent form; 10. For female subjects of childbearing age, the serum pregnancy test should be negative within 3 days before receiving the first dose (cycle 1, day 1).

Exclusion Criteria:

1. Have locally advanced unresectable or metastatic disease; unresectable includes unresectable stage III non-small cell lung cancer as defined by the Multidisciplinary Diagnosis and Treatment Consensus (2019 edition), including partial stages IIIA and IIIB and all stage IIIC, N2: single station mediastinal lymph nodes with short diameter≥3cm or N2: multi-station mediastinal metastasis with lymph node fusion and the short diameter of lymph node ≥2cm on CT, T4 invading esophagus, heart, aorta, pulmonary veins and all the N3;
2. NSCLC involving superior sulcus, large cell neuroendocrine carcinoma (LCNEC), sarcomatoid tumor;
3. Participants with known EGFR sensitive mutations or ALK translocation, EGFR and ALK mutation status needs to be identified for the subjects with non-squamous cell carcinoma;
4. Previous treatment with systemic antitumor therapy for early NSCLC, including investigational product;
5. History of (non-infectious) pneumonitis/interstitial lung disease requiring steroid treatment, or ongoing pneumonitis/interstitial lung disease requiring steroid treatment;
6. Active tuberculosis；
7. Active infection requiring systemic treatment；
8. Subjects with any known or suspected autoimmune disorder or immunodeficiency, with the following exceptions: hypothyroidism, hormone therapy is not needed, or well controlled at physiological dose; controlled type I diabetes;
9. Uncontrolled active hepatitis B (defined as positive hepatitis B surface antigen [HBsAg] in screening period with HBV-DNA detected higher than the upper limit of normal at the clinical laboratory of the study center); (the subjects with HBV-DNA assay <500 IU/mL within 28 days prior to randomization who have received local standard antiviral therapy for at least 14 days and are willing to receive antiviral therapy continuously during the study can be enrolled); active hepatitis C (defined as positive hepatitis C surface antibody [HCsAb] in screening period and positive HCV-RNA);
10. Known human immunodeficiency virus (HIV) infection (known positive HIV antibody);
11. Vaccination of live vaccine within 30 days prior to the first dose. Including but not limited to the following: parotitis, rubella, measles, varicella/ herpes zoster (varicella), yellow fever, Rabies, Bacille Calmette-Guérin (BCG) and typhoid vaccine (inactivated virus vaccine allowed);
12. ≥ grade 2 peripheral neuropathy；
13. Previous use of PD-1/PD-L1 agent or the drug acting on another targeted T cell receptor (e.g., CTLA-4, OX-40);
14. Severe allergic reaction to other monoclonal antibodies;
15. History of serious allergy to Pemetrexed, paclitaxel or docetaxel, cisplatin, carboplatin or its preventive medications;
16. Known serious or uncontrolled pre-existing diseases; including but not limited to cardiovascular events with hemodynamic instability, symptomatic cerebrovascular events, and hepatic cirrhosis above Child-Pugh A within 6 months;
17. History or current evidence of any disease, therapy or abnormal laboratory examination that may confuse the study results, interfere with subject's participation in the full course of the study or not meet the best interest of subject's participation in the study, as judged by investigators;
18. Other malignant tumors within 5 years prior to the first dose, except non-small cell lung cancer. The malignant tumors with negligible risk of metastasis or death (e.g., expected disease-free survival > 5 years) and expected to achieve radical outcomes after treatment (e.g., sufficiently treated carcinoma in situ of cervix, basal or squamous cell skin cancer, ductal carcinoma in situ treated for radical surgery) can be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 478 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
2-year Event Free Survival Rate | 2 years
  Event Free Survival (EFS):EFS is defined as the time from randomization until radiographic disease progression, local progression precluding surgery, inability to resect the tumor, local or distant recurrence, or death due to any cause. EFS determined either by biopsy assessed by central pathologist or by imaging using RECIST 1.1 assessed by BICR.
pCR rate | up to 7 weeks after neoadjuvant
  Pathological Complete Response (pCR) Rate :pCR rate is defined as the percentage of participants having an absence of residual invasive cancer in resected lung specimens and lymph nodes following completion of neoadjuvant therapy.

SECONDARY OUTCOMES:
Major Pathological Response | up to 7 weeks after neoadjuvant
  Major Pathological Response (mPR) Rate.mPR rate is defined as the percentage of participants having ≤10% viable tumor cells in the resected primary tumor and all resected lymph nodes in neoadjuvant therapy
Lymph node downstaging rate | up to 7 weeks after neoadjuvant
Perioperative complications | 90 days after the last administration
Treatment associated adverse events | 90 days after the last administration
  Adverse event (AE), abnormal laboratory examination, serious adverse event (SAE) related with the study drug judged using NCI-CTCAE V5.0; surgical feasibility: percentage of procedure delay or cancellation, change of surgical approach, operation time
EFS | up to 3 years
  EFS is defined as the time from randomization until radiographic disease progression, local progression precluding surgery, inability to resect the tumor, local or distant recurrence, or death due to any cause. EFS determined either by biopsy assessed by central pathologist or by imaging using RECIST 1.1 assessed by investigator
Disease-free survival (DFS) | up to 3 years
  DFS is defined as the time from postoperation until radiographic disease progression, , local or distant recurrence, or death due to any cause
Overall survival (OS) | up to 3 years
  OS is defined as the time from randomization until death from any cause.
R0 resection rate | up to 7 weeks after neoadjuvant
Surgical Completion Rate | up to 7 weeks after neoadjuvant

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
yes